CLINICAL TRIAL: NCT04787250
Title: Randomized Open Label, Parallel Group, Controlled Study to Evaluate the Safety and Surgery Sparing Effect of Phage Therapy With Antibiotics for Patients With Prosthetic Joint Infections Who Are Candidates for Two Stage Exchange Arthroplasty
Brief Title: Bacteriophage Therapy in Patients With Prosthetic Joint Infections
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Changes to protocol design
Sponsor: Adaptive Phage Therapeutics, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APT.PJI.001
Record Dates: First submitted 2021-02-18; First posted 2021-03-08 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Prosthetic Joint Infection
Keywords: Prosthetic; Joint; Knee; Hip; Phage; Bacteriophage; Prosthetic Joint
MeSH Terms: interventions — Phage Therapy; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: randomized, open-label, parallel-group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1, Phage Therapy with Antibiotic Treatment (Experimental): Phage therapy will be administered in conjunction with antibiotic treatment.
  Interventions: Biological: Phage Therapy
- Arm 2, Standard of Care (Active Comparator): Two-stage exchange arthroplasty entails resection arthroplasty and placement of an antibiotic-loaded spacer, antibiotic therapy, an antibiotic-free observation period, and re-implantation of a new prosthesis.
  Interventions: Procedure: Two-Stage Exchange Arthroplasty

INTERVENTIONS:
Biological: Phage Therapy — Phage will be administered based on patient's matching results.
  Other Names: Antibiotics
  Arms: Arm 1, Phage Therapy with Antibiotic Treatment
Procedure: Two-Stage Exchange Arthroplasty — Performed per the study center's standard of care. No investigational products are used.
  Other Names: Antibiotics
  Arms: Arm 2, Standard of Care

SUMMARY:
This is a study designed to evaluate bacteriophage therapy in patients with chronic prosthetic joint infections.

DETAILED DESCRIPTION:
This is a study designed to evaluate bacteriophage therapy in patients with chronic prosthetic joint infections of the hip or knee caused by 1 or 2 of the following organisms: Staphylococcus aureus, Staphylococcus epidermidis, Staphylococcus lugdunensis, Streptococcus sp., Enterococcus faecium, Enterococcus faecalis, Escherichia coli, Pseudomonas aeruginosa, and/or Klebsiella pneumoniae.

This study will also compare the safety and efficacy of phage therapy in conjunction with antibiotics versus standard of care (SOC) two-stage exchange arthroplasty plus antibiotics.

ELIGIBILITY:
General Inclusion Criteria:

* Males or females ≥18 years of age.
* Female patients of childbearing potential who agree to use contraception.
* Candidate for a two-stage exchange arthroplasty.
* Chronic prosthetic joint infection

General Exclusion Criteria:

* Prior history of prosthetic joint infections (PJI) of same joint treated surgically other than one prior Debridement Antibiotics and Implant Retention procedure
* Soft tissue defect requiring reconstruction
* Hardware misalignment or loosening
* Active osteomyelitis
* Septic shock or hemodynamic instability
* Stage 4 or greater chronic kidney disease
* Liver disease
* Decompensated cirrhosis
* Alcohol abuse or alcohol induced liver disease or non-alcoholic steatohepatitis
* Decompensated heart failure
* Any other clinically significant disease, per judgement of the investigator
* Neutropenia (neutrophil count < 1000 cells/cubic mm), thrombocytopenia (platelets < 50,000/cubic mm) or aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) > 3 time the upper limit of normal
* HIV, hepatitis C, hepatitis B infection
* Positive drug screen
* Receipt of chemotherapy, immunosuppressants or immune modulators
* Anti-viral medication
* Any known phage allergy
* Breast feeding or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of phage therapy | Day 1 through Week 26
  Incidence and type of adverse events and infusion reactions

SECONDARY OUTCOMES:
Efficacy of phage therapy to prevent need for surgery in patients with hip/knee prosthetic joint infections. | 6 weeks after completion of phage therapy
  Proportion of phage-treated patients with no need for surgery by no evidence of a prosthetic joint infection.
Efficacy of phage therapy in hip joint functionality as assessed by hip disability and osteoarthritis outcome questionnaire score (HOOS). | Week 26
  Time to reach minimum clinically important difference in hip dysfunction and osteoarthritis outcome score.
Efficacy of phage therapy in knee joint functionality as assessed by knee injury and osteoarthritis outcome questionnaire score (KOOS). | Week 26
  Time to reach minimum clinically important difference in knee injury and osteoarthritis outcome score.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hopkins, MD, Study Director — Adaptive Phage Therapeutics
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No